CLINICAL TRIAL: NCT02661152
Title: DAHANCA 30: A Randomized Non-inferiority Trial of Hypoxia-profile Guided Hypoxic Modification With Nimorazole During Radiotherapy/Chemoradiotherapy of Squamous Cell Carcinoma of the Head and Neck.
Brief Title: DAHANCA 30: A Randomized Non-inferiority Trial of Hypoxia-profile Guided Hypoxic Modification of Radiotherapy of HNSCC.
Acronym: DAHANCA30
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Head and Neck Cancer Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DAHANCA 30
Record Dates: First submitted 2016-01-14; First posted 2016-01-22 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Radiotherapy; Hypoxic Modification; Hypoxia; Gene Profile, Gene Signature
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypoxia | interventions — Nimorazole

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radio-/Chemoradiotherapy + nimorazole (Experimental): Hypoxia profile guided non-responder (less hypoxic tumour) to nimorazole but receiving the drug, which is normal standard radiotherapy of HNSCC in Denmark.
  Interventions: Drug: Nimorazole
- Radio-/Chemoradiotherapy (No Intervention): Hypoxia profile guided non-responder (less hypoxic tumour) to nimorazole and not receiving the drug, that is normally part of standard radiotherapy of HNSCC in Denmark.

INTERVENTIONS:
Drug: Nimorazole — Hypoxia gene profile is expected to discriminate between HNSCC responders and non-responders to hypoxic modification with nimorazole during radiotherapy. In DAHANCA 30 expected non-responders are randomized to +/- nimorazole during radiotherapy (non-inferiority study). Thus, similar efficacy of radiotherapy is expected in these groups. More hypoxic tumours receive nimorazole after DAHANCA standards.
  Arms: Radio-/Chemoradiotherapy + nimorazole

SUMMARY:
Hypoxic modification of radiotherapy with nimorazole has previously been shown to increase radiosensitivity in hypoxic head and neck squamous cell carcinomas (HNSCC).

In Denmark, nimorazole is added the radiotherapy of most HNSCC, as it has not previously been possible to discriminate more hypoxic tumours from less hypoxic tumours.

A hypoxia gene profile has shown to discriminate between responders and non-responders to nimorazole.

In DAHANCA 30, expected hypoxia profile guided non-responders are randomized to +/- nimorazole during radiotherapy.This in order to verify clinical use of the gene profile in selecting the relevant patients for hypoxic modification of radiotherapy with nimorazole.

DETAILED DESCRIPTION:
Hypoxic modification of radiotherapy with nimorazole has in the DAHANCA 5 trial been shown to increase radiosensitivity in hypoxic head and neck squamous cell carcinomas (HNSCC).

Previously, it has not been possible to discriminate more hypoxic tumours from less hypoxic tumours. Thus, nimorazole has been added the radiotherapy of most HNSCC.

Recently, a hypoxia gene profile has been developed, that discriminate between more and less hypoxic tumours. The basis of the discrimination is the cumulated expression of 15 hypoxia responsive genes, quantified from the tumour biopsy.

The profile has been validated on the independent DAHANCA 5 cohort. There was a significant effect of adding nimorazole to the radiotherapy of more hypoxic tumours as estimated with the gene profile, whereas there was no effect of adding nimorazole to the less hypoxic tumours. In a test for interaction, there was a significantly different response to nimorazole in the more hypoxic tumours compared to the less hypoxic tumours.

In the Dahanca 30 trial it is aimed to verify, that there is no benefit of supplying the radiotherapy of less hypoxic HNSCC with nimorazole. Thus, to explore whether it is possible to avoid the sideeffects of nimorazole without risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck squamous cell carcinoma with indication for hypoxic modification with nimorazole in accordance to the Danish Head and Neck Cancer guidelines (DAHANCA guidelines).
* Informed consent

Exclusion Criteria:

* Previous or present malignant disease conflicting with the radiotherapy treatment or evaluation of the treatment.
* Participation in a conflicting protocol.
* Initiation of radiotherapy more than 3 weeks after inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1252 (Estimated)
Dates: Start 2016-09; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with locoregional tumour control | 5 years
  Patients are being followed with regular clinical examinations for 5 years after therapy. Side effects, tumour control and survival status is registered in the DAHANCA database. Interim analysis are planned every 12 months.

SECONDARY OUTCOMES:
Number of participants with disease specific survival | 5 years
  Patients are being followed with regular clinical examinations for 5 years after therapy. Side effects, tumour control and survival status is registered in the DAHANCA database. Interim analysis are planned every 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, MD DMSc, Study Chair — DAHANCA Danish Head and Neck Group
Locations (1):
- Department of Experimental Clinical Oncology, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No